CLINICAL TRIAL: NCT03401983
Title: Effectiveness of Pelvic Floor Muscle and Abdominal Training in Women With Stress Urinary Incontinence: A Randomized Controlled Study
Brief Title: Effectiveness of Pelvic Floor Muscle and Abdominal Training in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hatice Kahyaoglu Sut, Head of Department of Obstetrics and Gynecology Nursing, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Effectiveness of Pelvic Floor
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Muscle Weakness
Keywords: exercise; pelvic floor; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PFMT + AT (Experimental): Pelvic Floor Muscle Training and Abdominal Training
  Interventions: Other: Pelvic Floor Muscle Training and Abdominal Training
- PFMT (Active Comparator): Pelvic Floor Muscle Training
  Interventions: Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Pelvic Floor Muscle Training and Abdominal Training — Pelvic Floor Muscle Training + Abdominal Training program was used in the study. The follow-up measurements of the PFMT+AT group were obtained in the 0th, 4th, and 8th weeks.
  Arms: PFMT + AT
Other: Pelvic Floor Muscle Training — Pelvic Floor Muscle Training program was used in the study. The follow-up measurements of the PFMT group were obtained in the 0th, 4th, and 8th weeks.
  Arms: PFMT

SUMMARY:
The aim of this study was to investigate the effectiveness of pelvic floor muscle and abdominal training in reproductive-age patients with stress urinary incontinence.

This prospective randomized controlled design study included 64 female patients aged 18-49 years with stress urinary incontinence. The patients were divided into 2 groups (32 PFMT "Pelvic Floor Muscle Training" and 32 PFMT+AT "Abdominal Training") by computer-based randomization. The stress urinary incontinence type was assessed by a stress test, and the pelvic floor muscle strength was measured with a home biofeedback device. Voiding functions were assessed by a 3-day voiding diary and uroflowmetric test. The UDI-6 scale was used to assess the urinary symptoms, and the IIQ-7 scale was used to assess the quality of life. The follow-up measurements of both groups were obtained in the 0th, 4th, and 8th weeks.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effectiveness of pelvic floor muscle and abdominal training in reproductive-age patients with stress urinary incontinence.

This prospective randomized controlled design study included 64 female patients aged 18-49 years with stress urinary incontinence. The patients were divided into 2 groups (32 PFMT "Pelvic Floor Muscle Training" and 32 PFMT+AT "Abdominal Training") by computer-based randomization. The stress urinary incontinence type was assessed by a stress test, and the pelvic floor muscle strength was measured with a home biofeedback device. Voiding functions were assessed by a 3-day voiding diary and uroflowmetric test. The UDI-6 scale was used to assess the urinary symptoms, and the IIQ-7 scale was used to assess the quality of life. The follow-up measurements of both groups were obtained in the 0th, 4th, and 8th weeks.

Participation of 29 patients from each group in the study was determined as sufficient to test the two-way hypothesis, with an effect size of 0.75, with an alpha level of 0.05, and with a power of 80%. However, 32 patients from each group were included as a precaution against possible missing data.

These women were randomly divided into the PFMT+AT (n=32) and PFMT (n=32) groups using a computer based randomization scheme. The data were collected from both groups at the 0th, 4th, and 8th weeks.

ELIGIBILITY:
Inclusion Criteria

* 18-49 years
* Meet the diagnosis of simple female stress urinary incontinence (Degree 0 or 1)
* Volunteer to participate the study

Exclusion Criteria

* BMI ≥30
* Hysterectomy, urinary incontinence or pelvic floor operations
* Chronic health problem (cardiovascular, cerebral, diabetes, liver, kidney, psychiatric disease, etc.)
* Urge urinary incontinence, mixed urinary incontinence, overflow urinary incontinence
* SUI Degree ≥2
* Symptomatic urinary tract infection
* During pregnancy or lactation period

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 64 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline pelvic floor muscle strength at 8 weeks | 0th, 4th, and 8th weeks.
  Pelvic floor muscle strength was measured using a perineometry device

SECONDARY OUTCOMES:
Change from baseline UDI-6 score at 8 weeks | 0th, 4th, and 8th weeks.
  Urinary symptoms were measured using the Urinary Distress Inventory (UDI-6)
Change from baseline IIQ-7 score at 8 weeks | 0th, 4th, and 8th weeks
  Urinary symptoms were measured using the Incontinence Impact Questionnaire (IIQ-7),

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322